CLINICAL TRIAL: NCT05768516
Title: Can we Improve Care Pathway in Low Back Pain? A Pilot Study
Brief Title: Can we Improve Care Pathway in Low Back Pain?
Acronym: DeltaDos
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Collaborators: Haute Ecole de Santé Vaud (Other); Delta SA (Unknown); University of Applied Sciences of Western Switzerland (Other); smarter medicine choosing wisely Switzerland (Unknown)
Responsible Party: Principal Investigator, Stephane Genevay, Professor, University Hospital, Geneva
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2023-00199
Record Dates: First submitted 2023-02-07; First posted 2023-03-14 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Back Pain, Low
Keywords: Stratified care; Guideline implementation; Primary care
MeSH Terms: conditions — Low Back Pain | interventions — Primary Health Care

STUDY DESIGN:
Intervention Model Description: Two-arms parallel pilot study. Two healthcare centres (one for each arm) have been selected for their convenience.
Who Masked: Outcomes Assessor
Masking Description: Participants and general practitioners will not be blinded to their group. No outcome will be measured be an external assessor (patients will fill out questionnaires at home). The statistical analysis will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-level intervention (Experimental): General practioners in this arm will receive the multi-level intervention composed of Stratified care, Healthcare professional education, Patient education and Interprofessional collaboration.
  Interventions: Other: Implementation of best practice for low back pain in primary care
- Usual care (No Intervention): GPs in the control group will have no specific training or intervention. They will treat patients according to their usual practice.

INTERVENTIONS:
Other: Implementation of best practice for low back pain in primary care — 1. Stratified care: GPs will use a simple algorithm based on the risk of chronicity to determine the management plan. The risk level bas will be based on the Start Back Tool (SBT) and other variables that have been shown to improve the classification, such as work capacity.
  2. Healthcare professional education: GPs will receive education to improve their knowledge about low back pain guidelines, diagnostic triage, patient education, stratified care and best practice.
  3. Patient education: An education booklet "Understanding My Low Back Pain" will be used by GPs during their consultations. Second, GPs, PTs and OTs will provide similar reassuring messages and direct patients to the website www.infomaldedos.ch.
  4. Interprofessional collaboration: A structured assessment form and a facilitated contact will be implemented between healthcare providers.
  Arms: Multi-level intervention

SUMMARY:
The general objective of this pilot study is to investigate a new multi-level intervention in primary care to improve the care of patients with low back pain. Specifically, it will first investigate the feasibility of delivering this intervention in primary care in Switzerland. Second, it will evaluate the effectiveness of the intervention on the use of unnecessary imaging and unhelpful medication in primary care, the risk of developing chronic disabling care, and direct and indirect healthcare costs.

In this two-arm parallel pilot study, it is the general practitioners that will be recruited to be in either arm. In the intervention group, they will deliver the multi-level intervention that consists of:

* Stratifying care based on the risk of chronicity
* Improving healthcare professional education
* Improving patient education
* Facilitating interprofessional communication

General practitioners in the control group will have no specific training or intervention. They will treat patients according to their usual practice.

DETAILED DESCRIPTION:
This study aims to investigate a multi-level intervention in primary care to improve the care of patients with LBP.

In this pilot trial, it is the GPs that will be recruited to be in either arm. Five to seven GPs will be recruited in each study arm. As this is a pilot study, randomization was not felt necessary. To facilitate this pilot study, two health care centers (one for each arm) have been selected for their convenience. GPs from each arm will thus be recruited within the same health care center.

For the development of the intervention, various existing interventions that have been tested successfully elsewhere and had the possibility of being adapted in the context of Switzerland's primary care practice were selected. The investigators used available evidence to develop the multi-level intervention. The different components and the procedures of the multi-level intervention were developed by a team of LBP experts in collaboration with GPs, PTs, and OTs. Various meetings with GPs were conducted to determine the feasibility and their preferences for each component of the intervention.

The overall goal of the intervention is to help GPs provide high-value care, adapt the treatment plan to the risk of chronicity (stratified care), decrease unnecessary healthcare (i.e., unnecessary imaging), and facilitate interprofessional collaboration. The intervention includes the following components:

1. Stratifying the management of LBP according to risk factors for chronicity with the StartBack tool (SBT) has been shown to improve patient outcomes and reduce unnecessary overtreatment. This stratification into 3 stages, low, medium, and high, is mainly based on the presence of elements such as kinesiophobia and catastrophism. These elements are linked to anxiety, which is often involved in the erroneous prescription of imaging or inappropriate care (e.g. opioids). Thus, by adapting management to psychological factors it is possible to facilitate the reduction of unnecessary care together with the improvement of patients' outcomes. Based on previous work, the investigators developed a simple algorithm to determine the risk level based on the SBT and other variables that have been shown to improve the classification, such as work capacity. Based on the risk level, a management plan is proposed which may include PT.

   PTs in the intervention group will all have participated to a one-day course to upgrade their knowledge on good clinical practice in LBP care and get the certification.
2. Healthcare professional education. The first component is health practitioners' education to improve their knowledge about LBP guidelines, diagnostic triage, and best practice. Furthermore, they will be trained to improve patients' education (i.e. on reducing the use of imaging), to follow a care strategy based on a questionnaire-based chronicity risk stratification rather than a step-up strategy, and improve interprofessional communication.
3. Patient education. Many patients expect to have an MRI of their spine in the belief that it will uncover the source of their problem and define the appropriate treatment. Only through better education can they change their perspective, be reassured of their clinical course without imaging, and understand the utility of staying active. Different strategies will be implemented to reassure patients. First, an education booklet "Understanding My Low Back Pain", which showed promising results in reducing the use of imaging has been translated into French and will be used by GPs during their consultations. Second, GPs, PTs, and OTs will provide similar reassuring messages and direct patients to the website www.infomaldedos.ch, which provides accurate and reassuring messages about LBP.
4. Interprofessional collaboration. By improving communication between the different healthcare providers, patients will have access to the right care at the right time and will receive a more consistent and reassuring message about LBP. To this end, a structured assessment form and facilitated contact will be implemented. PTs and OTs will be trained to provide a simple structured report of the patient's progress with a suggestion for further management to the GPs.

The multi-level intervention will be only at the level of the GPs. Prior to the start of the study, GPs will be informed on all aspects of good clinical practice during a specific time dedicated to continuing medical education. This will be done in interactive sessions, starting from their own experience, and implementing specific information when needed. A clinical pathway according to the risk of chronicity and specifically adapted to the Swiss healthcare system will be discussed during two one-hour meetings. The education will be provided by a rheumatologist with internationally recognized experience in the management of LBP. An information meeting will then be held to explain in detail the mechanisms of the study and the different tools that will be provided.

At the time of patient's first consultation for a new episode of back pain, The GP will have access to an interactive specifically designed and validated booklet in French "Understanding My Low Back Pain" to help educate patients that imaging is not recommended and point towards the general principle of good clinical practice care.

After the medical consultation, When the patient returns the signed informed consent form, the medical assistant will tag the patient within the computer system. Five days after the medical consultation the patient will receive an email with a questionnaire including the SBT. GPs will receive via email a summary of the SBT indicating the risk of chronicity (low, medium, or high) and a proposed treatment approach based on stratified care. The risk assessment will be based on the validated SBT with the addition of the ability to work.

In the case of low-risk GP'a are encouraged to focus on information and reassurance, with the help of information on a website. The use of additional treatments should be reduced to a minimum. In the case of medium risk, the proposition will be to prescribe 6 individual sessions of exercise-based physiotherapy. At the end of the 6 sessions, the physiotherapist will provide the GP with a structured report of the patient's progress with a suggestion for further management based on the clinical course: end of treatment, continuation for a few more sessions, or referral for further assessment to consider the need for structured multidisciplinary intervention. In cases of high risk, patients will be referred for 1-2 sessions to a specifically trained occupational therapist to determine if there is a need for immediate integration in a structured multidisciplinary group intervention or if the patient can be treated according to the proposition for medium risk patients. GPs are free to organize the following appointment and treatment plan according to the proposition or not.

Six weeks later, a second email will be sent to the patients with the same set of questionnaires and the updated results, including the updated risk of chronicity, will be sent to the GPs again. GPs may use this information to adapt patient care.

During the entire process, the decision on how to treat the patients is in the hand of the treating GPs. It is his responsibility to follow the recommendation of the proposed clinical pathway or not.

GPs in the control group will have no specific training or intervention. They will treat patients according to their usual practice. The same information will be provided to patients in the informed consent form (i.e. participation in a study on back pain). Patients will receive the same SMS to verify their phone number and then receive the same questionnaire as in the "stratified care" group. However, no feedback will be provided to the GPs.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18
* Patient consulting a general practitioner for a new episode of LBP
* Patients is part of "Delta Network"

Exclusion Criteria:

* Patients that had already consulted their GP for LBP in the last three months (not a new episode)
* Patients unable to give consent and/or unable to answer the questionnaires, i.e. due to Dementia or language difficulties
* Known pregnancy
* Unable or unwilling to provide either a smartphone number or an email address.
* Unable or unwilling to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of imaging and opioids prescriptions | At 6 months
  The number of imaging procedure and opioids prescription in each group will be calculated
Recruitment procedures | At 6 months
  The number of patients included in the pilot trial in a 6-month period (number of participants/month/GP)

SECONDARY OUTCOMES:
Level of disabling low back pain (LBP) | At 6 weeks, 3 months and 6 months
  The level of disabling LBP will be measured with the Core Outcome Measure Index (COMI)
Percentage of LBP patients reaching "acceptable symptom states " | At 6 weeks, 3 months and 6 months
  the number of patients reaching the "patient acceptable symptom state" (PASS) level as defined on the Core Outcome Measure Index (COMI)
Level of low back pain intensity | At 6 weeks, 3 months and 6 months
  The level of low back pain intensity will be measured with the Numerical rating scale (NRS) pain scale. This scale is from 0 to 10 (higher score equals to higher pain intensity).
Percentage of patients reaching a low level of low back pain intensity | At 6 weeks, 3 months and 6 months
  The level of low back pain intensity will be measured with the Numerical rating scale (NRS) pain scale from 0 to 10. A low level is defined as equal or inferior to 2.0.
Global perceived change | At 6 weeks, 3 months and 6 months
  Global perceived change (GPC) by the patient on a 6 points Likert scale ranging from "fully recovered" to "much worse"
Low back pain trajectory | At 6 months
  Percentage of patients in each category according to low back pain trajectories
Direct treatment costs of low back pain | At 6 months
  The direct treatment costs of LBP will be divided in several categories: GP visits, Specialists visit, pain medication, physiotherapy and investigations (blood tests and imaging studies)
Working incapacity costs | At 6 months
  The working incapacity costs will be calculated based on the answers given in the Work Productivity and Activity Impairment Questionnaire (WPAI)
Beliefs about low back pain in healthcare practitioners | At 6 months
  Beliefs about low back pain will be evaluated in healthcare practitioners at the end of the intervention to identify the presence of unhelpful beliefs with the Back Pain Attitude Questionnaire (Back-PAQ).

OTHER OUTCOMES:
Age | enrollment
  Age
Sex | enrollment
  Sex
Body mass index | enrollment
  Body mass index
Comorbidities | enrollment
  The presence of comorbidities will be evaluated at the start of the study
Tobacco use | enrollment
  Tobacco use will be evaluated at the start of the study

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Genevay, Prof, Principal Investigator — University Hospital, Geneva
Locations (2):
- Switzerland (2):
  - Centre médical Lignon, Le Lignon, Canton of Geneva
  - Centre médical Onex, Onex, Canton of Geneva

IPD SHARING:
Plan to Share IPD: No
Anonymized data will be made available on request.